CLINICAL TRIAL: NCT00629447
Title: A Pilot Trial of Innohep (Tinzaparin) Low Molecular Weight Heparin for Primary Prophylaxis of Venous Thromboembolism in Brain Tumor Patients
Brief Title: Innohep for Prophylaxis of Venous Thromboembolism in Brain Tumor Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00008486; 4930 (Other: Duke Legacy IRB Number)
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Primary Brain Tumor
Keywords: Primary Brain Tumor; Venous Thromboembolism; Heparin
MeSH Terms: conditions — Brain Neoplasms; Venous Thromboembolism | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The patients will receive a single daily subcutaneous injection of Tinzaparin at 4500 IU.
  Interventions: Drug: Innohep

INTERVENTIONS:
Drug: Innohep — The patients will receive a single daily subcutaneous injection of Tinzaparin at 4500 IU.
  Other Names: Tinzaparin

SUMMARY:
To determine the safety of prophylaxis with Tinzaparin low molecular weight heparin in primary brain tumor patients. 2. To determine the incidence of deep venous thrombosis or pulmonary embolism in brain tumor patients who will be receiving Tinzaparin as primary prophylaxis. 3. To determine the overall survival of patients with malignant glioma who receive Tinzaparin. 4. To determine the bone density before and after prophylactic Tinzaparin.

DETAILED DESCRIPTION:
Many patients with brain tumors develop thinning of the bones and weak bones, called osteoporosis. At baseline (or within 4 weeks of enrollment onto study) and 12 months the subject will have a bone densitometry study (DEXA-Scan) which is a test to determine bone density (the measure of the strength and thickness of bones) by using x-ray techniques.

A single arm pilot trial will be performed with newly diagnosed pathologically confirmed malignant glioma patients. The patients will receive low molecular weight heparin (Tinzaparin), which will begin at least 48 hours after craniotomy or stereotactic biopsy, but no later than four weeks after the most recent surgery.

The patients will receive a single daily subcutaneous injection of Tinzaparin at 4500 IU.

The primary analysis will be conducted at six months and the safety will be determined by the incidence of clinically significant bleeding, ≥ grade III/IV CNS hemorrhage or grade II hemorrhage elsewhere. The Tinzaparin will be discontinued for any grade II or higher hemorrhage, except CNS hemorrhage and patients with asymptomatic CNS hemorrhage seen on a scan (grade III) at study entry will stay on Tinzaparin, except if the CNS hemorrhage expands or there is a new hemorrhage, in which case the Tinzaparin will be discontinued. For patients without a CNS hemorrhage at entry, a new asymptomatic CNS hemorrhage (grade III), or a CNS hemorrhage with symptoms (≥ grade IV) will result in discontinuation of the Tinzaparin. If the patient does not have any hemorrhage, the Tinzaparin will be continued for an additional six months with the second analysis performed at 12 months. Patients may stay on Innohep as long as they are benefiting and there are no adverse reactions necessitation stopping therapy. Patients will continue to having the same labs and clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed pathologically confirmed WHO Grade III or Grade IV glioma (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed glioma, gliosarcoma and glioblastoma multiforme);
2. Patients must be 18 years of age or older at the time of informed consent;
3. Karnofsky performance status 60% and a life expectancy of at least 6 months;
4. The patient is at least 48 hours after craniotomy or stereotactic biopsy but no later than four weeks from the last surgical procedure;
5. Adequate hematologic function as demonstrated by laboratory values performed within 14 days: platelet count > 100,000, prothrombin time (PT) 1.2 x control, inactivated partial thromboplastin time (aPTT) 1.2 x control;
6. Signed informed consent prior to patient registration.

Exclusion Criteria:

1. Presence of a coagulopathy, as defined by laboratory parameters including a platelet count < 100,000, PT > 1.2 x control or a PTT > 1.2 x control.
2. Symptomatic intracranial bleeding, which includes inter- or intratumor bleeding and causes mass effect or neurological disability control;
3. The presence of acute or chronic deep venous thrombosis demonstrated by ultrasonography or venography. A baseline screening ultrasound or venogram is not required;
4. Active systemic bleeding, such as gastrointestinal bleeding or gross hematuria;
5. Excessive risk of bleeding as defined by stroke within the prior 6 months, history of CNS or intraocular bleed, or septic endocarditis;
6. Prior history of documented DVT or PE;
7. History of immune mediated heparin induced thrombocytopenia, as documented by a platelet count < 50,000 and positive heparin-induced platelet aggregation test;
8. Contraindication to tinzaparin or other heparins, including allergy or hypersensitivity to heparin or pork products, sulfite allergy, benzyl alcohol allergy or have or had had an epidural catheter or traumatic spinal puncture within 7 days prior to screening;
9. Serum creatinine >3.0 mg/dl;
10. Patient or partner of childbearing potential and not using adequate contraception;
11. Pregnant or nursing (women of childbearing potential may have a screening pregnancy test at the discretion of the investigator);
12. Medical condition requiring long-term anticoagulants such as atrial fibrillation or a mechanical heart valve;
13. Inability to give informed consent;
14. Inability to comply with study procedures, including subcutaneous injections and diagnostic procedures;
15. Participating in another study of an investigational agent at the time of enrollment. The use of an experimental or investigational regimen of an approved product is not cause for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Neurologic evaluation, CBC, Coagulation test (PT w/ INR, aPTT),Karnofsky performance status, Thrombosis panel, Adverse events assessment | MONTHS 2, 4, 6, 9, 12

SECONDARY OUTCOMES:
Bone densitometry study (DEXA-Scan)d | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James Vredenburgh, MD, Principal Investigator — Duke University Heatlh Systems
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States